CLINICAL TRIAL: NCT03879408
Title: Randomized, Double-Blind, Placebo And Active Controlled, Study To Evaluate Two Strengths Of Concomitantly Dosed Naproxen Sodium With Acetaminophen, Compared With Naproxen Sodium and Hydrocodone/Acetaminophen In Postoperative Dental Pain
Brief Title: Naproxen Sodium/Acetaminophen Proof of Concept Dosing Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSPAA001068
Record Dates: First submitted 2019-03-01; First posted 2019-03-18 (Actual); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Pain
Keywords: Analgesics; Dental Pain; Naproxen; Acetaminophen; Pain
MeSH Terms: conditions — Pain; Toothache | interventions — Naproxen; Acetaminophen; Hydrocodone

STUDY DESIGN:
Intervention Model Description: Post-operative dental pain following third molar extraction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 440 mg naproxen sodium with 1000 mg acetaminophen (Experimental): 440 mg naproxen sodium with 1000 mg acetaminophen administered as a single dose of two naproxen sodium 220 mg tablets and two acetaminophen 500 mg tablets
  Interventions: Drug: 440 mg naproxen sodium with 1000 mg acetaminophen
- 220 mg naproxen sodium with 650 mg acetaminophen (Experimental): 220 mg naproxen sodium with 650 mg acetaminophen administered as a single dose of one naproxen sodium 220 mg tablet and two acetaminophen 325 mg tablets and one placebo tablet
  Interventions: Drug: 220 mg naproxen sodium with 650 mg acetaminophen
- 10 mg hydrocodone + 650 mg acetaminophen (Active Comparator): 10 mg hydrocodone + 650 mg acetaminophen administered as a single dose of two hydrocodone 5 mg + acetaminophen 325 mg tablets and two placebo tablets
  Interventions: Drug: 10 mg hydrocodone + 650 mg acetaminophen
- 440 mg naproxen sodium (Active Comparator): 440 mg naproxen sodium administered as a single dose of two naproxen sodium 220 mg tablets and two placebo tablets
  Interventions: Drug: 440 mg naproxen sodium
- Placebo tablet (Placebo Comparator): Single dose of four placebo tablets
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 440 mg naproxen sodium with 1000 mg acetaminophen — 440 mg naproxen sodium with 1000 mg acetaminophen administered as a single dose of two naproxen sodium 220 mg tablets and two acetaminophen 500 mg tablets
  Other Names: Naproxen Sodium with Acetaminophen - High Dose
  Arms: 440 mg naproxen sodium with 1000 mg acetaminophen
Drug: 220 mg naproxen sodium with 650 mg acetaminophen — 220 mg naproxen sodium with 650 mg acetaminophen administered as a single dose of one naproxen sodium 220 mg tablet and two acetaminophen 325 mg tablets and one placebo tablet
  Other Names: Naproxen Sodium with Acetaminophen - Low Dose
  Arms: 220 mg naproxen sodium with 650 mg acetaminophen
Drug: 10 mg hydrocodone + 650 mg acetaminophen — 10 mg hydrocodone with 650 mg acetaminophen administered as a single dose of two hydrocodone 5 mg + acetaminophen 325 mg tablets and two placebo tablets
  Other Names: Commercial Hydrocodone + Acetaminophen Tablet
  Arms: 10 mg hydrocodone + 650 mg acetaminophen
Drug: 440 mg naproxen sodium — 440 mg naproxen sodium administered as a single dose of two naproxen sodium 220 mg tablets and two placebo tablets
  Other Names: Naproxen sodium
  Arms: 440 mg naproxen sodium
Drug: Placebo tablet — Single dose of four placebo tablets
  Arms: Placebo tablet

SUMMARY:
Study assessing efficacy and safety of concomitantly dosed naproxen sodium with acetaminophen, compared with naproxen sodium, hydrocodone/acetaminophen and Placebo in a postoperative dental pain.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo- and active-controlled, parallel-group study to evaluate the analgesic efficacy and safety of concomitantly administered naproxen sodium 440 mg with acetaminophen 1000 mg and concomitantly administered naproxen sodium 220 mg with acetaminophen 650 mg, compared with a fixed combination of hydrocodone 10 mg/acetaminophen 650 mg, naproxen sodium 440 mg, and placebo over a twelve-hour period after surgical extraction of four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. Males of females 17-50 years old
2. Weigh 100 pounds or greater and have a body mass index (BMI) of 18.5 to 35 (inclusive) at screening
3. Surgical removal of up to four third molars, of which, two must be mandibular impactions
4. Meets requirements for post -surgical pain level
5. Females of childbearing potential and males agree to contraceptive requirements of study
6. Have a negative urine drug screen at screening, and on day of surgical procedure

Exclusion Criteria:

1. Pregnant female, breastfeeding, trying to become pregnant or male with pregnant partner or partner currently trying to become pregnant
2. Have known allergy or hypersensitivity to naproxen or other NSAIDS, including aspirin, or to acetaminophen, tramadol, hydrocodone or other opioids
3. Not able to swallow large tablets or capsules
4. History of any condition (s) in investigator's opinion, may jeopardize subject safety, well-being and integrity of study
5. Use analgesics 5 or more times per week
6. History of chronic tranquilizer use, heavy drinking, substance abuse as judged by investigator site staff within last 5 years
7. Use of immunosuppressive drugs within 2 weeks of screening
8. History of peptic ulcer disease or gastrointestinal bleeding in the last two years or hematologic bleeding

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 290 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — Jean Brown Research (JBR)
Locations (1):
- Jean Brown Research Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Placebo: Participants received a single oral dose of four placebo tablets at baseline (Day of surgery-Day 1).
- Arm 2: Naproxen Sodium 440 mg: Participants received a single oral dose of naproxen sodium 440 milligrams (mg)(administered as two naproxen sodium 220 mg tablets) and two placebo tablets at baseline (Day of surgery-Day 1).
- Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg: Participants received a single oral dose of naproxen sodium 220 mg tablet (administered as one naproxen sodium 220 mg tablet) and acetaminophen 650 mg (two acetaminophen 325 mg tablets) and one placebo tablet at baseline (Day of surgery-Day 1).
- Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg: Participants received a single oral dose of naproxen sodium 440 mg (administered as two naproxen sodium 220 mg tablets) and acetaminophen 1000 mg (two acetaminophen 500 mg tablets) at baseline (Day of surgery-Day 1).
- Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg: Participants received a single oral dose of hydrocodone 10 mg (administered as two hydrocodone 5 mg tablets) and acetaminophen 650 mg (two acetaminophen 325 mg tablets) and two placebo tablets at baseline (Day of surgery-Day 1).
Period: Overall Study
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Started | 35 | 69 | 61 | 63 | 62
Completed | 33 | 65 | 58 | 62 | 61
Not Completed | 2 | 4 | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg | Total
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (1.50) | 19.0 (2.39) | 18.2 (1.33) | 19.0 (2.23) | 18.3 (1.70) | 18.6 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 36 | 33 | 35 | 32 | 155
  Male | 16 | 33 | 28 | 28 | 30 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 5 | 6 | 6 | 34
  Not Hispanic or Latino | 27 | 60 | 56 | 57 | 56 | 256
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 1 | 4
  Asian | 0 | 3 | 2 | 4 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 | 2 | 0 | 6
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  White | 32 | 61 | 57 | 54 | 57 | 261
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Sum of Pain Intensity Difference Score From Baseline (0 Hour) to 6 Hours (SPID 0-6)
Description: Time-weighted sum of the pain intensity difference (SPID) score was measured using a Pain Intensity-Numerical Rating Scale (PI-NRS) ranging from 0-10 (0 = no pain, 10 = very severe pain). The possible range of SPID for 0-6 hours was from -60 to 60. A higher value of SPID indicated greater pain relief. PID was the difference between baseline pain intensity and pain intensity at assessment. Time-weighted sum of the pain intensity difference scores were derived by first multiplying each PID score by the time from the previous time point and adding these time-weighted PID scores together over the intervals from 0 to 6 hours.
Time Frame: Baseline (0 hour) up to 6 hours post-dose
Population: Intent-to-Treat (ITT) analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 2.36 (2.181) | 25.59 (1.562) | 30.28 (1.677) | 33.77 (1.633) | 23.60 (1.651)

2. Primary Outcome: Time-weighted Sum of Pain Intensity Difference Score From Baseline (0 Hour) to 12 Hours (SPID 0-12)
Description: Time-weighted sum of the pain intensity difference score was measured using a PI-NRS ranging from 0-10 (0 = no pain, 10 = very severe pain). The possible range of SPID for 0-12 hours was from -120 to 120. A higher value of SPID indicated greater pain relief. PID was the difference between baseline pain intensity and pain intensity at assessment (12 hours). Time-weighted sum of the pain intensity difference scores were derived by first multiplying each PID score by the time from the previous time point and adding these time-weighted PID scores together over the intervals from 0 to 12 hours.
Time Frame: Baseline (0 hour) up to 12 hours post-dose
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 5.80 (4.666) | 50.07 (3.341) | 55.47 (3.587) | 66.43 (3.494) | 39.94 (3.533)

3. Secondary Outcome: Time-Weighted Sum of Total Pain Relief Score From Baseline (0 Hour) to 6 Hours (TOTPAR 0-6)
Description: Time-weighted total pain relief (TOTPAR) was measured using a Pain Relief Numerical Rating Scale (PR-NRS) ranging from 0-10 (0 = no relief, 10 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value was 0, and the maximum value was 60. Higher scores was indicative of more pain relief.
Time Frame: Baseline (0 hour) up to 6 hours post-dose
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 7.96 (2.581) | 35.20 (1.848) | 40.94 (1.984) | 45.13 (1.933) | 32.88 (1.954)

4. Secondary Outcome: Time-Weighted Sum of Total Pain Relief Score From Baseline (0 Hour) to 8 Hours (TOTPAR 0-8)
Description: TOTPAR was measured using a PR-NRS ranging from 0-10 (0 = no relief, 10 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value was 0, and the maximum value was 80. Higher scores was indicative of more pain relief.
Time Frame: Baseline (0 hour) up to 8 hours post-dose
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 11.12 (3.554) | 47.19 (2.545) | 54.37 (2.732) | 60.78 (2.662) | 41.61 (2.691)

5. Secondary Outcome: Time-Weighted Sum of Total Pain Relief Score From Baseline (0 Hour) to 12 Hours (TOTPAR 0-12)
Description: TOTPAR was measured using a PR-NRS ranging from 0-10 (0 = no relief, 10 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value was 0, and the maximum value was 120. Higher scores was indicative of more pain relief.
Time Frame: Baseline (0 hour) up to 12 hours post-dose
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 18.20 (5.595) | 69.96 (4.006) | 76.80 (4.301) | 90.22 (4.190) | 57.03 (4.237)

6. Secondary Outcome: Time-Weighted Sum of Pain Intensity Difference Score From Baseline (0 Hour) to 8 Hours (SPID 0-8)
Description: Time-weighted sum of the pain intensity difference score was measured using a PI-NRS ranging from 0-10 (0 = no pain, 10 = very severe pain). The possible range of SPID for 0-8 hours was from -80 to 80. A higher value of SPID indicated greater pain relief. PID was the difference between baseline pain intensity and pain intensity at assessment (8 hours). Time-weighted sum of the pain intensity difference scores were derived by first multiplying each PID score by the time from the previous time point and adding these time-weighted PID scores together over the intervals from 0 to 8 hours.
Time Frame: Baseline (0 hour) up to 8 hours post-dose
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale | 3.24 (2.981) | 34.11 (2.134) | 39.98 (2.291) | 45.27 (2.232) | 29.58 (2.257)

7. Secondary Outcome: Pain Relief (PAR) Scores at Individual Timepoints
Description: Participants answered a question at individual time points: "how much relief do you have from your starting pain?" on a 11-point PR-NRS. Scale ranged from 0=no relief to 10=complete relief. Higher score indicated improvement in pain.
Time Frame: 0.25 hours, 0.5 hours, 0.75 hours, 1 hours, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours, and 12 hours
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale
  0.25 hours | 0.45 (0.26) | 0.80 (0.18) | 1.36 (0.20) | 1.07 (0.19) | 1.04 (0.20)
  0.5 Hours | 0.51 (0.44) | 2.27 (0.31) | 3.46 (0.33) | 4.03 (0.33) | 3.23 (0.36)
  0.75 Hours | 0.77 (0.48) | 4.11 (0.35) | 5.10 (0.37) | 5.71 (0.36) | 5.08 (0.36)
  1 Hours | 1.06 (0.49) | 5.29 (0.35) | 5.91 (0.38) | 6.60 (0.37) | 6.03 (0.37)
  1.25 Hours | 1.13 (0.49) | 5.99 (0.35) | 6.46 (0.38) | 7.17 (0.37) | 6.40 (0.37)
  1.5 Hours | 1.18 (0.48) | 6.36 (0.34) | 6.89 (0.37) | 7.65 (0.36) | 6.44 (0.36)
  2 Hours | 1.08 (0.48) | 6.62 (0.34) | 7.37 (0.37) | 7.97 (0.36) | 6.38 (0.36)
  3 Hours | 1.37 (0.49) | 6.52 (0.35) | 7.61 (0.38) | 8.24 (0.37) | 6.26 (0.37)
  4 Hours | 1.66 (0.51) | 1.46 (0.36) | 7.68 (0.39) | 8.46 (0.38) | 5.96 (0.38)
  5 Hours | 1.59 (0.52) | 6.45 (0.37) | 7.43 (0.40) | 8.23 (0.39) | 5.54 (0.40)
  6 Hours | 1.53 (0.53) | 6.26 (0.38) | 7.23 (0.41) | 8.15 (0.40) | 4.88 (0.40)
  7 Hours | 1.51 (0.55) | 6.05 (0.39) | 6.80 (0.42) | 7.94 (0.41) | 4.50 (0.41)
  8 Hours | 1.65 (0.54) | 5.95 (0.39) | 6.63 (0.42) | 7.71 (0.41) | 4.23 (0.41)
  9 Hours | 1.61 (0.56) | 5.73 (0.40) | 6.27 (0.43) | 7.44 (0.42) | 3.88 (0.43)
  10 Hours | 1.73 (0.58) | 5.71 (0.42) | 5.66 (0.45) | 7.49 (0.44) | 3.66 (0.44)
  11 Hours | 1.86 (0.60) | 5.71 (0.43) | 5.33 (0.46) | 7.26 (0.45) | 3.91 (0.46)
  12 Hours | 1.89 (0.61) | 5.62 (0.44) | 5.18 (0.47) | 7.25 (0.46) | 3.98 (0.46)

8. Secondary Outcome: Pain Intensity Difference (PID) Scores at Individual Time Points
Description: Pain Intensity was self-reported over 12 hours, using a pain rating of 0-10 on the PI-NRS, with score ranged from 0-10 (0= no pain; 10 = worst imaginable pain). Pain intensity differences were calculated with respect to baseline at each time point after study drug administration.
Time Frame: as for outcome 7
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 61 | 63 | 62
Units on a scale
  0.25 hours | 0.25 (0.21) | 0.58 (0.15) | 1.01 (0.16) | 0.85 (0.15) | 00.79 (0.16)
  0.5 Hours | 0.07 (0.33) | 1.82 (0.24) | 2.61 (0.25) | 3.06 (0.25) | 2.36 (0.25)
  0.75 Hours | 0.24 (0.38) | 3.15 (0.27) | 3.82 (0.29) | 4.31 (0.29) | 3.77 (0.29)
  1 Hours | 0.45 (0.39) | 3.97 (0.28) | 4.41 (0.30) | 4.95 (0.29) | 4.48 (0.30)
  1.25 Hours | 0.34 (0.40) | 4.50 (0.28) | 4.87 (0.30) | 5.42 (0.30) | 4.71 (0.30)
  1.5 Hours | 0.31 (0.39) | 4.72 (0.28) | 5.18 (0.30) | 5.76 (0.29) | 4.74 (0.30)
  2 Hours | 0.22 (0.40) | 4.87 (0.28) | 5.49 (0.31) | 6.01 (0.30) | 4.67 (0.30)
  3 Hours | 0.34 (0.41) | 4.75 (0.30) | 5.62 (0.32) | 6.17 (0.31) | 4.51 (0.31)
  4 Hours | 0.53 (0.43) | 4.63 (0.31) | 5.64 (0.33) | 6.31 (0.32) | 4.26 (0.33)
  5 Hours | 0.50 (0.44) | 4.59 (0.32) | 5.51 (0.34) | 6.13 (0.33) | 3.89 (0.34)
  6 Hours | 0.47 (0.44) | 4.50 (0.32) | 5.28 (0.34) | 6.06 (0.33) | 3.39 (0.34)
  7 Hours | 0.40 (0.45) | 4.36 (0.32) | 4.96 (0.34) | 5.82 (0.34) | 3.08 (0.34)
  8 Hours | 0.48 (0.45) | 4.17 (0.32) | 4.74 (0.34) | 5.68 (0.34) | 2.90 (0.34)
  9 Hours | 0.53 (0.46) | 4.04 (0.33) | 4.46 (0.35) | 5.41 (0.34) | 2.56 (0.35)
  10 Hours | 0.64 (0.40) | 4.01 (0.35) | 3.87 (0.37) | 5.43 (0.36) | 2.42 (0.37)
  11 Hours | 0.69 (0.50) | 3.99 (0.35) | 3.63 (0.38) | 5.16 (0.37) | 2.71 (0.37)
  12 Hours | 0.71 (0.50) | 3.91 (0.36) | 3.53 (0.38) | 5.16 (0.37) | 2.66 (0.38)

9. Secondary Outcome: Participant's Global Evaluation of Study Medication OR Overall Impression of Study Medication According to Participant's Global Evaluation
Description: Participants were asked to rate their overall impression of the study medication using the following scale: poor (0), fair (1), good (2), very good (3), and excellent (4) where higher score represented better outcome.
Time Frame: Up to 12 hours
Population: ITT analysis set included all randomized participants. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
Number analyzed (Participants) | 35 | 69 | 60 | 63 | 61
Units on a Scale | 0.8 (0.18) | 2.7 (0.13) | 2.9 (0.14) | 3.3 (0.13) | 2.7 (0.14)

ADVERSE EVENTS:
Time Frame: Up to Day 10
Description: The safety analysis set included all participants who were randomized and took investigational product.
Arm/Group | Arm 1: Placebo | Arm 2: Naproxen Sodium 440 mg | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/69 | 0/61 | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/69 | 0/61 | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 14/35 | 5/69 | 8/61 | 9/63 | 22/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Placebo (N=35) | Arm 2: Naproxen Sodium 440 mg (N=69) | Arm 3: Naproxen Sodium 220 mg + Acetaminophen 650 mg (N=61) | Arm 4: Naproxen Sodium 440 mg + Acetaminophen 1000 mg (N=63) | Arm 5: Hydrocodone 10 mg + Acetaminophen 650 mg (N=62)
Nausea (Gastrointestinal disorders) | 9 | 2 | 2 | 3 | 20
Vomiting (Gastrointestinal disorders) | 7 | 2 | 4 | 6 | 9
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Alveolar osteitis (Infections and infestations) | 0 | 1 | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 1 | 3
Headache (Nervous system disorders) | 4 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03879408/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03879408/SAP_001.pdf